CLINICAL TRIAL: NCT00328250
Title: Internet Insomnia Intervention: Development and Feasibility
Brief Title: Effectiveness of Internet Cognitive Behavioral Therapy Intervention for Treating Insomnia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lee M Ritterband, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12232; R34MH070805 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Internet; CBT; Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive the online CBT intervention immediately and will use the online program for 8 weeks
  Interventions: Behavioral: Cognitive behavioral treatment (CBT) delivered over the Internet
- 2 (Active Comparator): Participants will receive the online CBT intervention after a 4-month waiting period
  Interventions: Behavioral: Cognitive behavioral treatment (CBT) delivered over the Internet

INTERVENTIONS:
Behavioral: Cognitive behavioral treatment (CBT) delivered over the Internet — CBT delivered over the Internet for insomnia targets maladaptive behaviors and dysfunctional thoughts that perpetuate sleep problems. Treatment includes through educational, behavioral, and cognitive strategies.

SUMMARY:
This study will evaluate the effectiveness of an online cognitive behavioral therapy intervention in improving sleep, mood, and cognitive functioning in people with insomnia.

DETAILED DESCRIPTION:
Insomnia is a disorder that is characterized by a perception or complaint of inadequate or poor-quality sleep. Symptoms of insomnia include difficulty falling asleep, waking frequently during the night and having difficulty returning to sleep, waking too early in the morning, and unrefreshing sleep. Insomnia may also cause problems during the day, such as tiredness, difficulty concentrating, and irritability. Cognitive behavior therapy (CBT) has been found to have significant short- and long-term benefits for people with insomnia. Access to CBT for many people, however, is limited, due to the high cost of treatment and a lack of trained professionals in some locations. Delivering CBT via the internet could help make the treatment more widely available. This study will evaluate the effectiveness of an online CBT intervention in improving sleep, mood, and cognitive functioning in people with insomnia.

Participants in this open label study will be randomly assigned to receive the online CBT intervention either immediately or after a 4-month waiting period. Participants will use the online program for 1 to 2 hours per week for 8 weeks. Participants will keep track of their sleep patterns for the first and last 2 weeks of a 4-month period by keeping a daily diary and wearing a wrist watch device that monitors movement. All participants will report to the study site for baseline evaluations before beginning treatment and for final evaluations upon completing the program, about 4 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Subjective complaints of poor sleep
* Difficulties falling and/or staying asleep (sleep onset latency and/or wake after sleep onset is greater than 30 minutes; sleep efficiency is less than 85%)
* Sleep difficulties at least 3 nights per week
* Sleep difficulties have persisted for more than 6 months
* At least one daytime problem due to poor sleep (e.g., fatigue, performance impairment, or mood disturbance)
* Daytime problems due to sleep disturbances cause marked distress or significant impairment in social or occupational functioning
* Has internet access

Exclusion Criteria:

* Presence of other sleep disorders (as evaluated by specific questions from structured interview) (e.g., sleep apnea, periodic leg movements while sleeping, or parasomnias)
* Significant psychological distress (including clinical depression and anxiety), as determined using the Beck Depression Inventory (BDI), STPI, Patient Health Questionnaire (PHQ), and clinical interview
* Substance use or medical condition that causes sleep problems
* Currently receiving psychological treatment
* Taking medications that have not been stabilized for the 3 months prior to study entry
* Regularly goes to sleep after 2am or wakes after 9am
* Shift worker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency, total sleep time, total wake time, sleep-onset latency, wake after sleep onset, and early morning awakening | Measured at baseline and Months 3 and 9
Insomnia Severity Index | Measured at baseline and Months 3 and 9
Beliefs and attitudes about sleep as measured by the Dysfunctional Beliefs and Attitudes about Sleep scale (DBAS 16) | Measured at baseline and Month 3
Sleep knowledge | Measured at baseline and Month 3
Fatigue as measured by the Multidimensional Fatigue Symptom Inventory (MFSI) | Measured at baseline and Month 3
Depression as measured by the Beck Depression Inventory 2 | Measured at baseline and Month 3
Anxiety as measured by the State-Trait Personality Inventory (STPI) | Measured at baseline and Month 3
Cognitive functioning as measured by the Headminder's Customized Research Tool (CRT) and Conner's Continuous Performance Test (CPT) | Measured at baseline and Month 3

SECONDARY OUTCOMES:
Cost-benefit measures (direct and indirect costs associated with insomnia) | Measured at baseline and Months 3 and 9
Quality of life as measured by the SF-12 Health Survey | Measured at baseline and Month 3
Feedback regarding use of the internet intervention, including post-treatment ratings of treatment credibility, acceptability, effectiveness, satisfaction, and ease of use of the internet | Measured at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Ritterband, PhD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Behavioral Health and Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Shaffer KM, Finkelstein EA, Camacho F, Ingersoll KS, Thorndike F, Ritterband LM. Effects of an Internet-Based Cognitive Behavioral Therapy for Insomnia Program on Work Productivity: A Secondary Analysis. Ann Behav Med. 2021 Jun 2;55(6):592-599. doi: 10.1093/abm/kaaa085. PMID 33057694
- [Derived] Shaffer KM, Hedeker D, Morin CM, Ingersoll K, Thorndike F, Ritterband LM. Intraindividual variability in sleep schedule: effects of an internet-based cognitive-behavioral therapy for insomnia program and its relation with symptom remission. Sleep. 2020 Dec 14;43(12):zsaa115. doi: 10.1093/sleep/zsaa115. PMID 32511726
- [Derived] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560